CLINICAL TRIAL: NCT02692066
Title: Response and Clearance of Viral DNA Following Administration of Live Attenuated Varicella Vaccine in Children With Liver Disease
Brief Title: Response and Clearance of Viral DNA Following Administration of Live Attenuated Varicella Vaccine.
Status: Withdrawn | Type: Observational
Why Stopped: Funding not acquired
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 15-2042
Record Dates: First submitted 2016-02-19; First posted 2016-02-25 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Varicella; Transplants
MeSH Terms: conditions — Chickenpox | interventions — Chickenpox Vaccine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Controls: Healthy Children ages 6 months-21 years who have not received varicella vaccine and who do not have prior varicella or zoster will receive Varivax. We will then measure 1) markers of humoral immunity at baseline and 4 weeks post vaccination and 2) markers of cell mediated immunity at baseline, 1 week, and 4 weeks post vaccination
  Interventions: Biological: varicella vaccine
- Children with Chronic Liver Disease: Children with chronic liver disease ages 6 months-21 years who have not received varicella vaccine and who do not have prior varicella or zoster will receive Varivax. We will then measure 1) varicella DNA in the blood and saliva at enrollment, 1 week, 2 weeks, 3 weeks, 4 weeks post vaccination 2)markers of humoral immunity at baseline and 4 weeks post vaccination and 3) markers of cell mediated immunity at baseline, 1 week, and 4 weeks post vaccination
  Interventions: Biological: varicella vaccine

INTERVENTIONS:
Biological: varicella vaccine

SUMMARY:
Varicella zoster virus (VZV) can lead to significant morbidity and mortality in transplant recipients. Current recommendations suggest a 4 week waiting period between vaccination and transplantation and consideration of booster immunizations if antibody response does not reach target levels. This four week waiting period can result in delayed transplant, rejection of an optimal organ, or missed opportunity to vaccinate. However, these recommendations are not evidence based.

This is a prospective study to look at the immune response to varicella vaccine in children with chronic liver disease.

Investigators will evaluate:

1. the time at which VZV DNA becomes undetectable in blood and saliva by PCR after vaccination in children with chronic liver disease and
2. the difference in humoral and cell mediated immune response to varicella immunization between children with chronic liver disease and healthy children.

ELIGIBILITY:
Inclusion Criteria:

* 6 months to 21 years
* no history of varicella, zoster or prior varicella vaccination

Exclusion Criteria:

* acute liver failure
* liver transplant anticipated within 28 days
* prior history of receiving blood products or immunoglobulin within 5 months prior to vaccination
* fever
* pregnancy
* immunocompromised status
* receiving immunosuppressive meds

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with liver disease and healthy controls who have not received varicella vaccination and who have no history of varicella or zoster
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Estimated); Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
clearance of viral DNA | 4 weeks
humoral response | 4 weeks
cell mediated response | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Amy Feldman, MD, Principal Investigator — University of Colorado, Denver